CLINICAL TRIAL: NCT00660517
Title: Randomized, Double-Blind Trial of MP29-02 Nasal Spray Compared to Placebo, Astelin Nasal Spray, and Fluticasone Propionate Nasal Spray in the Treatment of Patients With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP4001
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — MP29-02; azelastine; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MP29-02 (Experimental): azelastine HCl 548 mcg / fluticasone propionate 200 mcg nasal spray
  Interventions: Drug: MP29-02
- azelastine Hcl 548 mcg (Active Comparator): azelastine Hcl 548 mcg nasal spray
  Interventions: Drug: azelastine Hcl
- fluticasone propionate 200 mcg (Active Comparator): fluticasone propionate 200 mcg nasal spray
  Interventions: Drug: fluticasone propionate
- placebo (Placebo Comparator): placebo nasal spray
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MP29-02 — azelastine HCl 548 mcg / fluticasone propionate 200 mcg nasal spray one spray per nostril twice a day
  Arms: MP29-02
Drug: azelastine Hcl — azelastine Hcl nasal spray one spray per nostril two times a day
  Other Names: Astelin
  Arms: azelastine Hcl 548 mcg
Drug: fluticasone propionate — fluticasone propionate 200 mcg nasal spray one spray per nostril two times a day
  Other Names: generic Flonase
  Arms: fluticasone propionate 200 mcg
Drug: placebo — placebo nasal spray one spray per nostril two times a day
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if two allergy medications (azelastine and fluticasone) are more effective than placebo or either medication alone (azelastine or fluticasone)

DETAILED DESCRIPTION:
This will be a Phase III, randomized, double-blind, parallel-group study in subjects with moderate-to-severe SAR. The study will be conducted at 8 investigational sites during the 2007-2008 Texas Mountain Cedar allergy season. After a 7-day Placebo Lead-In Period (Day -7 to Day 1), subjects will be instructed to take placebo lead-in medication twice daily (1 spray per nostril), approximately every 12 hours. On Day 1, subjects who satisfy the symptom severity requirements and continue to meet all of the study inclusion/exclusion criteria will be randomized in a 1:1:1:1 ratio to receive 1 spray per nostril twice daily of MP29-02, azelastine hydrochloride, fluticasone propionate, or placebo nasal spray.

Efficacy will be assessed by the change from baseline in the subject-reported 12-hour reflective Total Nasal Symptom Score (TNSS), consisting of the sum of the scores of sneezing, nasal congestion, runny nose, and nasal itching. On Days -7 through 14, subjects will rate the TNSS symptoms, the TOSS symptoms of itchy eyes, watery eyes and eye redness, and the symptom of postnasal drip twice daily (AM and PM) in a diary prior to the dose of study medication. Symptoms will be scored on a 0 to 3 scale (0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms), such that the maximum daily symptom severity score will be 24 for the TNSS and 18 for the TOSS. The 12-hour reflective TNSS, the instantaneous TNSS, the 12-hour reflective score for postnasal drip, the 12-hour reflective TOSS, and the instantaneous TOSS will be calculated based on these scores. Additional secondary efficacy variables will include reflective and individual nasal and ocular symptom scores and change from Baseline to Day 14 in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ).

Subjects ≥ 18 years of age will complete the adult RQLQ on Day 1 (prior to dosing) and Day 14. Subjects will return to the clinic on Day 7 for an interim evaluation. After completing the 2-week double-blind treatment period, subjects will return to the clinic on Day 14 (or at time of early termination) for an end-of-study evaluation. Safety and tolerability assessments will be made on Days 7 and 14. Tolerability will be evaluated by subject reported adverse events (AEs), nasal examinations, and vital signs assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 12 years of age and older with a 2 year history of moderate to severe seasonal allergic rhinitis
* Must be in generally good health
* Must meet minimum symptom requirements, as specified in the protocol.
* Must be willing and able to provide informed consent and to participate in all study procedures
* Positive skin test to a prevalent Texas Mountain Cedar allergen

Exclusion Criteria:

* On Focused Nasal Examination, the presence of any nasal mucosal erosion, nasal ulceration, or nasal septal perforation (Grade 1b - 4) at either the screening visit or randomization visit will disqualify the subject from the study.
* Other nasal disease(s) likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa, clinically significant polyposis, or nasal structural abnormalities.
* Nasal surgery or sinus surgery within the previous year.
* Chronic sinusitis - more than 3 episodes per year
* Planned travel outside of the study area during the study period
* The use of any investigational drug within 30 days prior to Day screening. No investigational products are permitted for use during the conduct of this study
* Presence of any hypersensitivity to drugs similar to azelastine hydrochloride or fluticasone propionate
* Women who are pregnant or nursing
* Women of childbearing potential who are not abstinent or not practicing a medically acceptable method of contraception* see section 6.1.1
* Respiratory Tract Infections within 14 days prior to Day screening
* Respiratory Tract Infections requiring antibiotic treatment 14 days prior to screening
* Asthma (with the exception of mild, intermittent asthma). Subjects with mild, intermittent asthma who only require short-acting inhaled bronchodilators (not more often than twice per week) and who do not have nocturnal awakening as a result of asthma are eligible for enrollment
* Significant pulmonary disease including COPD
* Clinically significant arrhythmia or symptomatic cardiac conditions
* A known history of alcohol or drug abuse within the last 2 years
* Existence of any surgical or medical condition or physical or laboratory findings, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug; that might significantly affect the subject's ability to complete this trial; or their safety in this trial.
* Clinically relevant abnormal physical findings within 1 week of randomization which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (7):
- United States (7):
  - Allergy and Asthma Associates, Austin, Texas
  - Central Texas Research, New Braunfels, Texas
  - Southwest Allergy and Asthma Center, P.A., San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy, Asthma Research Center, San Antonio, Texas
  - Allergy and Asthma Care, Waco, Texas
  - Allergy and Asthma Center, Waco, Texas

REFERENCES:
- [Derived] Hampel FC, Ratner PH, Van Bavel J, Amar NJ, Daftary P, Wheeler W, Sacks H. Double-blind, placebo-controlled study of azelastine and fluticasone in a single nasal spray delivery device. Ann Allergy Asthma Immunol. 2010 Aug;105(2):168-73. doi: 10.1016/j.anai.2010.06.008. PMID 20674829

RESULTS

PARTICIPANT FLOW:
Groups:
- Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg: azelastine Hcl/ fluticasone propionate nasal spray one spray per nostril two times a day
- Azelastine Hcl 548 Mcg: azelastine Hcl nasal spray one spray per nostril two times a day
- Fluticasone Propionate 200 Mcg: fluticasone propionate nasal spray one spray per nostril two times a day
- Placebo: nasal spray
Period: Overall Study
Arm/Group | Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg | Azelastine Hcl 548 Mcg | Fluticasone Propionate 200 Mcg | Placebo
Started | 153 | 152 | 151 | 151
Completed | 145 | 144 | 144 | 144
Not Completed | 8 | 8 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg | Azelastine Hcl 548 Mcg | Fluticasone Propionate 200 Mcg | Placebo | Total
Number analyzed (Participants) | 153 | 152 | 151 | 151 | 607
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 11 | 10 | 13 | 43
  Between 18 and 65 years | 136 | 132 | 137 | 131 | 536
  >=65 years | 8 | 9 | 4 | 7 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (14.2) | 39.5 (14.1) | 38.1 (14.2) | 39.9 (14.7) | 39.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 97 | 100 | 102 | 396
  Male | 56 | 55 | 51 | 49 | 211
Region of Enrollment [Number; unit: participants]
  United States | 153 | 152 | 151 | 151 | 607

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12 Hour Reflective Total Nasal Symptom Score (rTNSS)
Description: change from baseline in the 12 hour reflective total nasal symptoms score(rTNSS) consisting of nasal congestion,runny nose,itchy nose and sneezing scored twice daily( AM and PM) in diary cards for the entire 14 day study period The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.
Time Frame: day 1 to day14
Population: Intent to Treat (ITT) population includes all subjects who were randomized and had at least one post baseline efficacy observation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg | Azelastine Hcl 548 Mcg | Fluticasone Propionate 200 Mcg | Placebo
Number analyzed (Participants) | 153 | 152 | 151 | 151
units on a scale | -5.3 (5.1) | -3.3 (4.2) | -3.8 (4.8) | -2.2 (4.2)

2. Secondary Outcome: Change From Baseline in 12 Hour Instantaneous Total Nasal Symptom Score (iTNSS)
Description: change from baseline in the 12 hour instantaneous total nasal symptoms score(iTNSS) consisting of nasal congestion,runny nose,itchy nose and sneezing scored twice daily( AM and PM) in diary cards for the entire 14 day study period.
  The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.
Time Frame: day 1 to day 14
Population: Intent to Treat (ITT) population includes all subjects who were randomized and had at least one post baseline efficacy evaluation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg | Azelastine Hcl 548 Mcg | Fluticasone Propionate 200 Mcg | Placebo
Number analyzed (Participants) | 153 | 152 | 151 | 150
units on a scale | -4.4 (5.2) | -3.0 (4.5) | -3.5 (4.8) | -1.7 (4.2)

3. Secondary Outcome: Change From Baseline in Adult ( Greater Than 18 Years of Age) Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)at the End of 14 Days
Description: Change from Baseline in adult ( greater than 18 years of age) Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)at the end of 14 days The measurement scale is 0 to 24. A reduction in symptom severity score is indicated by a negative value.
Time Frame: day 1 to day 14
Population: Intent to Treat(ITT) population (18 years of age or older) who have had at least one post baseline efficacy evaluation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg | Azelastine Hcl 548 Mcg | Fluticasone Propionate 200 Mcg | Placebo
Number analyzed (Participants) | 135 | 133 | 132 | 126
units on a scale | -1.6 (1.4) | -1.2 (1.3) | -1.4 (1.4) | -1.0 (1.3)

ADVERSE EVENTS:
Arm/Group | Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg | Azelastine Hcl 548 Mcg | Fluticasone Propionate 200 Mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/152 | 0/151 | 0/151
Other Adverse Events (participants affected / at risk) | 28/153 | 15/152 | 13/151 | 10/151
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelastine HCl 548 Mcg / Fluticasone Propionate 200 Mcg (N=153) | Azelastine Hcl 548 Mcg (N=152) | Fluticasone Propionate 200 Mcg (N=151) | Placebo (N=151)
dysgusia (Gastrointestinal disorders) | 11 (11) | 3 (3) | 0 (0) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 6 (6) | 5 (5)
headache (Nervous system disorders) | 4 (4) | 2 (2) | 6 (6) | 2 (2)
pharyngolaryngeal pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
acute sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators participating in multicenter studies must agree not to present data gathered individually or by a subgroup of centers before the full, initial publication, unless this has been agreed to by all other investigators and Meda Pharmaceuticals.

Meda Pharmaceuticals requests that it receive copies of any intended communication reasonably in advance (at least 15 working days for an abstract or oral presentation and 45 working days for a manuscript)